CLINICAL TRIAL: NCT03690531
Title: Efficacy of Mindfulness as an Intervention in the Pediatric Emergency Department
Status: Completed | Type: Observational
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Manager, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Other Study IDs: 2018-05-04
Record Dates: First submitted 2018-09-21; First posted 2018-10-01 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2018-09

CONDITIONS: Anxiety Fear; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Take Pause Virtual Reality Head Set: The mbVR intervention arm will be a Take-Pause virtual reality simulation will be for 5 minutes shown through a virtual reality goggle, headset and iPhone.
  Interventions: Device: Take-Pause virtual reality
- Passive Distraction Group_IPAD: The Passive Distraction group will utilize the standard or passive distraction technique of using an IPAD lasting 5 minutes.
  Interventions: Device: Passive Distraction

INTERVENTIONS:
Device: Take-Pause virtual reality — Take-Pause virtual reality simulation lasting 3 minutes shown through a virtual reality goggle, headset and iPhone.
  Groups: Take Pause Virtual Reality Head Set
Device: Passive Distraction — Standard or passive distraction technique, lasting 5 minutes.
  Groups: Passive Distraction Group_IPAD

SUMMARY:
Non-pharmacological interventions including distraction techniques (ie., games, ipads, bubbles, stickers) are standard of care in reducing situation anxiety for children in the pediatric emergency department. The goal of the study is to evaluate the efficacy of a mindfulness based virtual reality (mbVR) tool (Take-Pause) for pediatric patients age > 12 years. The study team will be providing children with a virtual reality experience upon arrival to the emergency department and measuring the effectiveness of the intervention versus standard of care (Ipads, games). Subjective measurements will include questionnaires and objective measurements will include vital signs.

DETAILED DESCRIPTION:
Emergency room visits can be a particularly stressful experience for children. It is well-known that among pediatric patients, increased anxiety and stress levels can contribute to less pain tolerance and higher pain scores. Increased levels of anxiety can also lead to difficulty communicating needs and building a good patient-provider relationship. Furthermore, higher situational anxiety may also lead to decreased patient satisfaction. Though there are pharmacologic interventions to mitigate pain and anxiety, the side effect profiles or route of administration sometimes outweigh the potential temporary benefits medication may provide. Distraction techniques have long been established in literature to help diminish pain in pediatric patients while essentially having no adverse profile. By utilizing a simple distraction such as visual or musical stimuli, providers have been able to decrease the use of anxiolytics or analgesics during pediatric care. Only a handful of controlled studies have explored distraction techniques in the pediatric emergency room, showing promising results in alleviating procedural pain/anxiety.

Immersive virtual reality has been introduced recently as an alternative distraction technique among hospitalized patients, providing a way to cope with the stressful hospital environment. Several randomized control studies have found virtual reality to significantly reduce pain in pediatric patients undergoing chronic or burn wound dressing changes. However, no studies have been done in the emergency room exploring the efficacy of virtual reality as a distraction technique, nor integrating mindfulness as part of the virtual reality experience. Mindfulness has garnered interest over the years as another powerful, but simple tool, in reducing emotional stress and increasing overall well-being of participants. An organization which has integrated mindfulness into a virtual reality program for adolescents is Take-Pause. The intervention will administer the Take-Pause immersive virtual reality simulation as a distraction technique via virtual reality goggles, headset, and iphone.

The study will be a prospective, single-blinded randomized control trial conducted in an pediatric emergency room at a single tertiary care hospital located in an urban region. The primary outcome is to decrease situational anxiety level by at least 5 points on a State Trait Anxiety Inventory scale when comparing mbVR to passive distraction technique. Secondary outcomes will look at reduction of perceived pain when utilizing the Wong-Baker FACES scale and respiratory rate or heart rate changes. Study population will consist of pediatric patients aged 13 to 17 year old presenting to the emergency room, enrolled during a 12 month period. Follow-up will be conducted at 5-min post-intervention. Exclusion criteria includes patients who have received opioid or anxiolytic pharmacologic intervention at triage or 1 hour prior to ED arrival. Patients will be randomly assigned after triage to either the mbVR or passive distraction intervention arm via a 1:1 patient allocation scheme utilizing block randomization. Baseline short STAI survey, pain scale, and vitals will be obtained during triage. The timer will begin once video starts and end when the video is complete. After 5 minutes, the patient will repeat the survey, scale, and have vitals taken. The treatment, or mbVR intervention arm will be a Take-Pause virtual reality simulation lasting 5 minutes shown through a virtual reality goggle, headset and iPhone. The control arm will consist of the standard or passive distraction technique, lasting 5 minutes. Each intervention arm will consist of 55 subjects for a total of 110 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the pediatric emergency room
* aged 13 years to 17 years
* understand and can complete instructions in English
* English-speaking.
* Participants must also be conscious and not in need of immediate interventions

Exclusion Criteria:

* Anxiolytic or opioid analgesic given in triage,
* developmental delay
* seizure
* significant visual impairment
* hearing impairment
* prone to motion sickness

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children between age 13 to 17 presenting to the emergency department
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Decrease in anxiety level | 5 minutes
  The primary outcome is to decrease situational anxiety level by at least 5 points on a State Trait Anxiety Inventory scale when comparing mbVR to passive distraction technique. The scores range from 20 to 80 with high score indicating higher levels of anxiety.

SECONDARY OUTCOMES:
Reduction in pain scores | 5 minutes
  Secondary outcomes will look at reduction of perceived pain when utilizing the Wong-Baker FACES scale ranges from 0 to 10 with 0 being no pain; 4-6 is moderate pain and 10 is severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: John Marshall, MD, Study Chair — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arane K, Behboudi A, Goldman RD. Virtual reality for pain and anxiety management in children. Can Fam Physician. 2017 Dec;63(12):932-934. PMID 29237632